CLINICAL TRIAL: NCT03512431
Title: Dose Adjustment of Tacrolimus Based on Home Sampling in Renal Transplant Recipients
Acronym: TacDrop
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Sandoz (Industry); The Norwegian association for renal disease and transplants (Unknown)
Responsible Party: Principal Investigator, Anders Åsberg, Head of Laboratory, Oslo University Hospital
Other Study IDs: TacDrop
Record Dates: First submitted 2018-04-10; First posted 2018-04-30 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Renal Transplant Rejection
Keywords: analytical method validation; renal transplantation; limited sampling strategy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood samples finger prick micro samples DNA extracted from venous whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Only one arm in the present study
  Interventions: Diagnostic Test: Micro sampling

INTERVENTIONS:
Diagnostic Test: Micro sampling — Compare finger prick micro samples with venous blood samples for measuring whole blood tacrolimus concentrations

SUMMARY:
Repeated 12-hour pharmacokinetic (PK) investigations in renal transplant recipients for parallel sampling of standard venous bloods samples and finger prick micro samples (Mitra tips). Primary aim to validate the micro sampling tacrolimus concentrations against venous blood concentrations.

DETAILED DESCRIPTION:
Renal transplant recipients using Prograf® as part of their immunosuppressive regimen will be included in the study. Patients will receive oral and written study information and sign the informed consent before entering the study. A 12-hour pharmacokinetic investigation will be performed when Tac doses have been stable for at least 7 days (approximately 3-4 weeks posttransplant). They will continue on unchanged doses of tacrolimus as before PK investigation 1 (PK1). After at least another 7 days a second 12h PK-investigation (PK2) will be performed. If Tac doses needs to be changed after PK1 and before PK2 the second PK will not be performed.

Tac doses and blood concentration obtained as part of standard follow-up of the patients will be included in a non-parametric population model to obtain individually optimal sampling times for each patient using the MMopt function in Pmetrics®. During both PK1 and PK2 the patients themselves will be instructed to take two "home sampling" micro samples (Mitra® microsampling device) just prior to the standard vacutainer samples are obtained. Both the micro- and vacutainer samples will be drawn in 2 parallel samples right after each other and one will be mailed to the laboratory via standard mail. During PK1 the sampling times will be the same and standardized for all patients; before (0h) and 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10 and 12 hours after dose administration. During PK2 individually optimized sampling times based on 2, 3 and 4 samples will be determined using the MMopt function in Pmetrics and utilizing all individual dose and concentration information from before PK2, including the rich sampling during PK1. Spread over the entire study period, at least 6 real life home samplings for trough (C0) of Tac will also be performed by the patient and mailed to the hospital.

Tacrolimus induced tremor will be measured with a center-developed method utilizing infrared determined positioning (sampling ever 5 ms) of hand joints in the x-, y, z axis.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients
* Females and males
* Patients receiving tacrolimus as part of their immunosuppressive therapy (clinical decision not influenced by this study)

Exclusion Criteria:

* Patients on concomitant drugs with known pharmacokinetic interaction with tacrolimus

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Renal transplant recipients in the first two months after transplantation
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Absolute bias of micro sample tacrolimus concentrations | Within one dose interval of 12 hours
  absolute bias (mico- minus vacutainer sampling) over the clinical range (1 to 40 µg/L) of micro sampled, including simulated "home sampled", Tac trough concentrations
Relative bias of micro sample tacrolimus concentrations | Within one dose interval of 12 hours
  Relative bias (mico- minus vacutainer sampling divided by vacutainer sampled) over the clinical range (1 to 40 µg/L) of micro sampled, including simulated "home sampled", Tac trough concentrations

SECONDARY OUTCOMES:
popPK Bayesian predicted tacrolimus trough concentration | Within one dose interval of 12 hours
  Absolute and relative predictive error of population pharmacokinetic Bayesian estimated Tac trough concentration based on LSS with 2, 3 and 4 individually optimal sampling times more than 2 hours from trough
PK Bayesian predicted tacrolimus AUC0-12 | Within one dose interval of 12 hours
  Absolute and relative predictive error of population pharmacokinetic Bayesian estimated Tac AUC0-12 based on LSS with 2, 3 and 4 individually optimal sampling times
Tacrolimus tremor PK/PD relation | Within one dose interval of 12 hours
  Description of the mathematical relation between measured tacrolimus blood concentrations and specific Tac tremor over a dose interval

CONTACTS AND LOCATIONS:
Overall Officials: Karsten Midtvedt, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital - Rikshospitalet, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No